CLINICAL TRIAL: NCT07399925
Title: Assessment of the Impact of Oral Health Training for Caregivers on the Oral Health-related Quality of Life of Residents in Nursing Homes
Acronym: EHPADENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Tours (Other); UNIVERSITY HOSPITAL, ORLEANS (Unknown); Centre Hospitalier Jacques Cœur - Bourges (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC25_0023
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Oral Health Training
Keywords: Nursing home; Aged; Quality of health care; Anxiety; Oral health training; Quality of life
MeSH Terms: conditions — Anxiety Disorders | interventions — Oral Health; Nursing Homes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residents / Caregivers group (Experimental): Caregivers : all staff providing oral care to residents (registered nurses, nursing assistants, medical-psychological assistants, hospital assistant service occupational therapists) Residents: mentally independent patients who have been residing in a nursing home for at least three months.
  Interventions: Other: Caregivers training in oral health in nursing homes

INTERVENTIONS:
Other: Caregivers training in oral health in nursing homes — Training for healthcare workers on oral hygiene and health in nursing homes will be organised around two modules.
  Modules will aim to improve/update the specific knowledge and skills required to provide oral care to dependent residents in order to reduce the level of anxiety that may be associated with it. To ensure that all caregivers have acquired the training content, an assessment will be carried out at the end of each module in the form of a quiz.
  At the end of this training course, a decision tree on 'Should I call the dentist?', summary sheets of the training course and protocol sheets will be made available in the various nursing homes to help maintain the knowledge acquired during the training and guide caregivers in organizing the care pathway.

SUMMARY:
With the ageing of the French population, the number of elderly people loosing their autonomy is increasing, leading to a growing need for care in residential establishments for dependent elderly people . For multiple reasons, the oral and dental health of the elderly is often when they're admitted to a nursing home (financiary issues, loss of mobility, cognitive impairement, etc.). It can continue to deteriorate after admission du to communication difficulties between care team and dentists. As these various constraints can limit the monitoring and management of the consequences of oral senescence, it is easy to understand the oral health deterioration in nursing home residents.

This worsening in oral health is all the more worrying because residents rarely express the need for care, until emergency. This lack of complaints calls for even greater vigilance. While general hygiene care is well carried out, the majority of nursing staff are uncomfortable with oral hygiene care, which sometimes end up neglected or insufficient. Among the reasons that could explain this lack of care, nursing homes staff often speak of a reluctance to carry them out, a lack of knowledge, or even a fear of investing in this oral sphere.

The purpose of this study is to demonstrate that nursing staff (nurse, orderlies, medical-psychological assistants and hospital service agents) oral health formation will help the development of knowledge and skills, and will improve the quality of life related to oral health of dependant people, while decreasing nursing staff anxiety levels in regards to dental care.

To this end, before and 6 months after training in oral hygiene care for carers, the quality of life in relation to the oral health of residents will be assessed using the GOHAI questionnaire. Caregivers' anxiety levels will be assessed using the STAI-Y questionnaire. At the end of the training, two caregivers will be designated as oral health referents in each nursing home and a support unit will be set up. Supporting documents to help make the decision to call the dentist and care protocols left on site will complete this system.

DETAILED DESCRIPTION:
Throughout life, the oral cavity plays a vital role in many essential functions such as chewing and social interactions (communication, smiling, etc.). Its ageing is accompanied by disturbances that affect the overall health and quality of life of elderly people, particularly when they are dependent and/or institutionalised.

In these frail patients, local changes (reduced salivary flow, presence of removable dentures, etc.) as well as general pathologies (diabetes, hypertension, etc.) and their treatments, combined with neglect of daily hygiene and a decline in immune defences, lead to an imbalance in the oral microbiome. This imbalance manifests itself in the accumulation of biofilm (dental plaque), weakening of oral tissues and a worsening of the overall clinical condition. This dysbiosis has consequences both at the somatic level (imbalance of diabetes, development of cardiovascular diseases, etc.) and in terms of patients' quality of life (eating disorders, pain, discomfort, communication difficulties).

To ensure a good quality of life in relation to oral health, daily care is therefore necessary to remove bacterial plaque and food debris from the teeth, mucous membranes and dentures.

With an ageing population, the number of seniors losing their independence is increasing and could reach nearly 4 million people by 2050. Faced with this demographic change, the increase in care needs in residential care homes for the elderly (EHPAD) is accompanied by a shift in patient profiles. Patients are increasingly older and increasingly dependent. They therefore require specific care that is both compassionate and respectful of residents.

Before entering nursing homes, elderly people face barriers to accessing conventional dental care (financial barriers, accessibility to practitioners). In addition, they generally have functional limitations such as physical mobility difficulties and cognitive impairments. As a result, the oral health of elderly people is often impaired by the time they are admitted to a care facility. Once these dependent individuals have entered care homes, communication difficulties between the care team and the dentist constitute an additional barrier to access to care. Thus, the fact that an elderly person is in an institution reduces their use of dental services by 25% compared to a population of elderly people living independently at home. Given these multiple constraints that can limit the monitoring and management of the consequences of ageing in the oral cavity, it is understandable that the oral health of institutionalised people in France is poor.

This oral deterioration is all the more worrying given that dependent patients rarely express their need for care until a dental emergency arises, such as pain, injury, infection or mobility issues. This lack of complaints calls for even greater vigilance on the part of healthcare staff. Oral and dental pathologies will thus be associated with silent disruptions to essential social functions such as phonation, diction and eating. This deterioration in quality of life leads dependent individuals into a vicious circle of social isolation. Combined with cognitive disorders, these disruptions can cause behaviours that complicate the care relationship (aggression, agitation, wandering or refusal of care).2 The integration of oral hygiene measures as part of comprehensive care tailored to the motor and cognitive specificities of nursing home residents therefore appears essential to maintaining their quality of life and 'ageing well and healthily'.

On a daily basis, residents in nursing homes are supported by qualified healthcare professionals: nurses, nursing assistants, medical-psychological assistants and hospital service agents acting as nursing assistants. A range of tools for assessing oral care needs are available to these non-dental healthcare professionals to guide them in their care of residents. However, the measurement qualities of these different tools appear uncertain. It is therefore understandable why their choice regarding care and treatment decisions for residents is guided primarily by the resident's quality of life. While general hygiene care is well provided, the majority of care staff are uncomfortable with oral care, which is sometimes neglected or insufficient (simple examination, and/or oral health education, and/or oral hygiene care). Among the reasons often cited to explain this lack of care are a reluctance to perform these tasks or a lack of knowledge. Faced with this care, which is considered complex and time-consuming, caregivers are calling for specific training and the implementation of protocols for oral cavity care.

Investigators hypothesise that training care workers in nursing homes in oral health will promote the development of knowledge and skills that will improve residents' quality of life in relation to their oral health.

In accordance of these, the purpose of this study is to demonstrate that nursing staff (nurse, orderlies, medical-psychological assistants and hospital service agents) oral health formation will help the development of knowledge and skills, and will improve the quality of life related to oral health of dependant people, while decreasing nursing staff anxiety levels in regards to dental care.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 65 or over.
* Are present in the facility.
* Are mentally independent (MMS score ≥ 20 assessed within the last 12 months).
* Consent participating the study, or who have obtained consent from a legal tutor where applicable.
* have been present full-time in the nursing home for at least 3 months.
* Speak and understand French.
* Have signed the non-objection form.

Exclusion Criteria:

* Those who are unable to understand or respond to the questionnaire.
* Those who are not affiliated with a social insurance.
* Those receiving palliative cares.
* Those who refuse oral hygiene cares.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Changes in the oral health-related quality of life of nursing home residents. | 6 months
  Measurement of oral health-related quality of life score, defined using the Geriatric Oral Health Assessment Index (GOHAI) before (D0) and 6 months after caregiver training (M6). In order to assess the link between this differential and the initial GOHAI score observed in the patient before the intervention, a linear regression model of the 'change-score model' type will be constructed after centring the variables.

SECONDARY OUTCOMES:
Healthcare professionals' anxiety levels changes | 6 months
  Comparison of anxiety levels among healthcare professionals as defined by the State-Trait Anxiety Inventory (Stai-Y) just before (D7) and 6 months after caregiver training (M6)
Alignment between training, training tools and the needs of caregivers. | During training for healthcare professionals on oral hygiene and oral health, between day 7 and day 30
  Assessment of training's suitability for healthcare professionals' needs immediately after training, using a self-administered questionnaire designed to assess the quality of the training's organisation and teaching methods, the level of satisfaction in terms of expectations, and the practical applicability of the training.
Changes in oral health care pathways for nursing home residents. | 6 months
  Oral healthcare pathways for nursing home residents will be defined based on oral healthcare referral and organisation procedures before (D0) and 6 months after caregiver's training (M6).
  The use of healthcare professionals involved in residents' oral care will be assessed through various referrals to healthcare facilities for oral care over the last 6 months (dentist, doctor, hospital or resident's refusal) and the organisation of the care pathway (resident, family, caregiver). These elements will be identified by interviewing residents and/or reviewing medical records.
Association between residents' quality of life related to oral health and caregivers' anxiety levels. | 6 months
  Relationship between quality of life in relation to oral health and the level of anxiety among caregivers will be approached by studying the correlation between the average differences between GOHAI and STAI-Y scores.
Association between residents' age at inclusion and variations in GOHAI | 6 months
  Association between the resident's age at inclusion and the variation in GOHAI will be assessed by implementing the residents' age into the regression model used to assess the primary objective.
Association between health-related quality of life at inclusion and variations in GOHAI. | 6 months
  The association between health-related quality of life at inclusion and variation in GOHAI will be assessed by implementing the quantitative measure of residents' health-related quality of life at inclusion into a regression model used to assess the primary objective.
  The quantitative measure of residents' overall health-related quality of life (EQ-VAS) will be derived from the EQ-5D-5L self-assessment of residents' health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No